CLINICAL TRIAL: NCT03351114
Title: Pilot Study Evaluating the Efficacy of a Topical PDE4 Inhibitor for Morphea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00086947
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Morphea
Keywords: Morphea, Localized Scleroderma
MeSH Terms: conditions — Scleroderma, Localized | interventions — crisaborole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Crisaborole 2% ointment (Experimental): Crisaborole 2% ointment applied to affected skin twice per day.
  Interventions: Drug: Crisaborole

INTERVENTIONS:
Drug: Crisaborole — Apply Crisaborole 2% ointment to affected skin twice per day.
  Other Names: Eucrisa

SUMMARY:
This is a pilot study to determine the safety and clinical efficacy of crisaborole 2% ointment in the treatment of morphea.

DETAILED DESCRIPTION:
A Phase 2, pilot, proof-of-concept, open label, single arm prospective study to assess the safety, tolerability and efficacy of using crisaborole 2% ointment for adult morphea. Patients identified by their physician, nurse, or other member of their clinical care team as meeting criteria for the study will be asked to apply crisaborole 2% ointment, twice daily, on affected plaques for 12 weeks. A 4 mm skin punch biopsy will be performed at baseline and at 12 weeks, on the same affected plaque. Dermal thickness will be measured and compared before and at the end of treatment. Patients will have a clinical assessment at baseline and at weeks 4, 8 and 12. After week 12, patients who need further treatment will undergo standard of care treatment as determined by their primary dermatologist. Physician and patient reported assessment and skin imaging will be performed at baseline, week 4, 8 and 12, and at week 20. Photography will also be performed at baseline and week 12. An optional post treatment follow-up will be performed at week 20.

Medication will be provided free of charge by Pfizer, as part of the grant that is funding this study. These will be dispensed by the study group at baseline and during the subsequent clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. >= 18 years of age
2. Clinical diagnosis of morphea.
3. <20% Total body surface area involvement.
4. Does not require systemic immunosuppressive therapy for morphea.
5. No immunosuppressive systemic therapy 1 month prior to starting the study (methotrexate, mycophenolate mofetil, azathioprine, cyclosporine, cyclophosphamide, prednisone >=10 mg PO daily).
6. No immunomodulating topical therapy (topical steroids or topical calcineurin inhibitor), and no topical vitamin D analogue, 2 weeks prior to starting study.
7. No allergy to crisaborole or vehicle.
8. No known renal disease
9. Able to give informed consent.

Exclusion Criteria:Subjects fulfilling any of the following criteria are not eligible for inclusion in this study.

1. Clinical diagnosis of depression or history of suicidal ideation.
2. Pregnant or breastfeeding women, with pregnant women being defined as the state of a female after conception until the termination of gestation, confirmed by a positive urine human chorionic gonadotropin (hCG) laboratory test. Women with a positive urine hCG at any time during the study will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adela Cardones, MD, Principal Investigator — Duke UMC
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crisaborole 2% Ointment
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Crisaborole 2% Ointment
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 51 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Reduction in Dermal Thickness of Sentinel Plaque
Description: Change in dermal thickness on skin biopsy. A sentinel plaque will be selected at baseline. A 4 mm skin punch biopsy will be performed at baseline and at 12 weeks, on the same affected plaque.
Time Frame: Baseline, 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole 2% Ointment
Number analyzed (Participants) | 7
Participants | 5

2. Secondary Outcome: Percentage of Reduction in DIET Score of Sentinel Plaque
Description: The DIET (Dyspigmentation, Induration, Erythema, and Telangiectasias) score is a physician-assessed, previously validated score. Range is 0-12, and a higher score denotes increased activity or severity.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of reduction
Arm/Group | Crisaborole 2% Ointment
Number analyzed (Participants) | 7
percentage of reduction | 33 (26)

3. Secondary Outcome: Percentage of Reduction in LoSCAT Score
Description: LoSCAT (Localized Scleroderma Cutaneous Assessment Tool ) score is a physician-assessed, previously validated score. It has 2 components, the LoSSI (localized scleroderma skin severity index, range 0-162), which measures disease activity, and LoSDI (localized scleroderma damage index, range 0-216). The higher the number, the higher the disease activity and damage, respectively.
Time Frame: Baseline,12 weeks
Measure: Mean (Standard Deviation); unit: percentage of reduction
Arm/Group | Crisaborole 2% Ointment
Number analyzed (Participants) | 7
percentage of reduction
  LoSSI (Activity) | 37.5 (29)
  LoSDI (Damage) | 5 (36)

4. Secondary Outcome: Percentage of Reduction in Skindex-29 Score
Description: Skindex-29 is a health-related quality of life score; minimum score 30, maximum 150. Lower score indicates a better quality of life.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of reduction
Arm/Group | Crisaborole 2% Ointment
Number analyzed (Participants) | 7
percentage of reduction | 25.7 (16.4)

5. Secondary Outcome: Change in Dermal Thickness of Sentinel Plaque by Ultrasonography
Description: B-Mode ultrasonographic imaging will be utilized to measure dermal thickness of the sentinel plaque
Time Frame: Baseline, 4, 8 and 12 weeks, optional at 20 weeks
Population: Data not collected.
Arm/Group | Crisaborole 2% Ointment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 weeks.
Arm/Group | Crisaborole 2% Ointment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT03351114/Prot_SAP_000.pdf